CLINICAL TRIAL: NCT06211712
Title: Efficacy and Safety of Human Urinary Kallidinogenase Combined With Endovascular Therapy in Acute Ischemic Stroke With Large Vessel Occlusion: A Prospective, Randomized, Double-blind, Placebo-controlled, Multi-center Study
Brief Title: Efficacy and Safety of Human Urinary Kallidinogenase Combined With Endovascular Therapy in Acute Ischemic Stroke With Large Vessel Occlusion
Acronym: HEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Collaborators: Shanghai Stroke Association (Unknown)
Responsible Party: Principal Investigator, Qiang Dong, Chief physician, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2023-707
Record Dates: First submitted 2023-12-28; First posted 2024-01-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Urinary Kallidinogenase (Experimental)
  Interventions: Drug: Experimental: Human Urinary Kallidinogenase
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator: Placebo

INTERVENTIONS:
Drug: Experimental: Human Urinary Kallidinogenase — Before the first day of endovascular therapy (non-bridging), dissolve Human Urinary Kallidinogenase in 100 mL 0.9% sodium chloride for intravenous injection, for the next 9 days, once a day for a total of 10 days.
  Arms: Human Urinary Kallidinogenase
Drug: Placebo Comparator: Placebo — Before the first day of endovascular therapy (non-bridging), dissolve placebo in 100 mL 0.9% sodium chloride for intravenous injection, for the next 9 days, once a day for a total of 10 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Human Urinary Kallidinogenase combined with endovascular therapy in acute ischemic stroke (AIS) patients with large vessel occlusion.

DETAILED DESCRIPTION:
A prospective, randomized, double-blind, placebo-controlled, multi-center study of Human Urinary Kallidinogenase or Placebo, combined with endovascular therapy for AIS patients with large vessel occlusion.

Approximately 120 eligible subjects will be randomized (1:1) to receive one of the following treatments for 10 days:

* Human Urinary Kallidinogenase combined with endovascular therapy (non-bridged)
* Placebo combined with endovascular therapy (non-bridged) Primary efficacy of Human Urinary Kallidinogenase will be evaluated at 90±7 days.

The safety of Human Urinary Kallidinogenase will be evaluated through 90±7 days.

End of study evaluation will occur at day 90±7 or premature discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Participant with acute anterior circulation ischemic stroke receiving endovascular treatment within 24 hours (non-bridged).
2. Age ≥18 years old.
3. The mRS score was 0-1 before onset.
4. ASPECT score of infarction on emergency CT ≥7.
5. Emergency CTA indicating AIS with large vessel occlusion (internal carotid artery, M1 or M2 segment of middle cerebral artery).
6. Emergency CTP or DWI suggesting infarct core body ≥10 mL and <100 mL, and low perfusion brain tissue volume/ infarct core volume> 1.2.
7. Participant is willing and able to comply with the study protocol, and sign the informed consent form (patient or surrogate).

Exclusion Criteria:

1. Participant with severe heart, liver and kidney dysfunction, coagulation dysfunction, intolerance to surgery, Human Urinary Kallidinogenase allergy, contrast agent allergy or other angiographic contraindications.
2. CT or MRI showed intracranial hemorrhagic diseases (such as hemorrhagic stroke, epidural hematoma, intracranial hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.).
3. Participant with previous cerebral hemorrhage, brain tumor, brain trauma or other brain diseases.
4. Taking ACEI antihypertensive drugs regularly and could not stop.
5. Participant with major surgery or severe trauma in the past 2 weeks.
6. Poor compliance and cannot fully follow the study protocol.
7. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ASPECT score evaluated using routine CT | on day 7 after EVT
Modified Rankin Scale (mRS) score | on day 90 after EVT

SECONDARY OUTCOMES:
Barthel index | on day 10 and 90 after EVT
Percentage of TIC ≥ 2b and mRS ≤2 | on day 90 after EVT
Changes of NIH Stroke Scale(NIHSS) score from baseline | day 1, 4, 7 and 10 after EVT
Changes of vital signs from baseline | day 1, 4, 7 and 10 after EVT
Changes of blood inflammatory index and vascular endothelial cell growth index from day 1 after EVT | day 7 after EVT
MRI and / or DWI examined | within 10 days to determine the infarct volume
Recurrence rate of ischemic stroke | within 90 days after EVT

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Dong, M.D., Principal Investigator — Huashan Hospital; Wenjie Cao, M.D., Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China